CLINICAL TRIAL: NCT05251298
Title: "Parkinson AKTIV - Non-pharmacological Treatments in an Innovative Parkinson's Network"- Evaluates the Efficacy of an Online Platform That Allows Neurologists and Therapists to Exchange Therapy Recommendations Regarding Their Patients With Parkinson's Disease (PwP), Communicate Assessments and Plan Physical Therapy, Occupational Therapy as Well as Speech and Swallowing Therapy
Brief Title: "Parkinson AKTIV - Non-pharmacological Treatments in an Innovative Parkinson's Network"
Acronym: ParkinsonAKTIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: privates Institut für angewandte Versorgungsforschung GmbH (Unknown); AOK PLUS (Industry)
Responsible Party: Principal Investigator, Dr. Tobias Warnecke, Professor Dr. Tobias Warnecke, University Hospital Muenster
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-356-f-S; 01NVF19002 (Other Grant/Funding Number: Gemeinsamer Bundesausschuss; Innovationsausschuss)
Record Dates: First submitted 2021-12-09; First posted 2022-02-22 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
Keywords: Activities of Daily Living; Disease Management; Quality of Life; Rehabilitation; Patient-Centered Care; Delivery of Health Care; Integrated Care
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Patients in the intervention group come from the same region (Münsterland) and will undergo therapies coordinated through the online platform.
  Interventions: Other: Coordination through the online platform "JamesAKTIV"
- Control group (No Intervention): Patients in the control group will undergo their usual therapies as prescribed by their neurologists.

INTERVENTIONS:
Other: Coordination through the online platform "JamesAKTIV" — Coordination of the treatment through the online platform "JamesAKTIV" that allows neurologists and therapists to select specialised therapies for the predominant symptoms of the patients and communicate easily about problems during the treatment
  Arms: Intervention group

SUMMARY:
The purpose of this study is to evaluate the efficacy of an online platform that allows neurologists and therapists to exchange therapy recommendations, communicate assessments and plan physical therapy, occupational therapy as well as speech and swallowing therapy for their patients.

DETAILED DESCRIPTION:
The aim of this study is to enroll 185 patients in the intervention group and 185 patients in the control group. Patients in the intervention group come from the same region (Münsterland), the control group will consist of patients outside this region. The patients in the intervention group undergo therapies planned and coordinated through the online platform for 12 months. The patients in the intervention group will be evaluated using the PDQ-39, UPDRS, H&Y as well as Schwab & England. The patients in the control group will be evaluated using the PDQ-39.

ELIGIBILITY:
Inclusion Criteria (Intervention Group):

* Idiopathic Parkinson's Disease with pharmacological treatment
* 30 years old or older
* place of residence: Münsterland, Tecklenburger Land, Kreis and Stadt Osnabrück
* sufficient knowledge of the German language, should be able to understand the consent form

Exclusion Criteria:

* severe cognitive deficits
* Atypical Parkinsonian Disorders
* participation in other studies

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2021-11-28 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life measured by PDQ 39 | Change from Baseline PDQ 39 at 12 months
  The Parkinson's Disease Questionnaire (PDQ-39, max. score of 100 indicates the worst quality of life)

SECONDARY OUTCOMES:
Change in Health-related resource use in the elderly population, assessed by FIMA | Change from Baseline FIMA at 12 months
  FIMA stands for "Questionnaire concerning Health-related resource use in the elderly population" and is a German questionnaire assessing the Health-related resource use in the elderly population
Change in disease severity measured by UPDRS | Change from Baseline UPDRS at 12 months
  UPDRS - Unified Parkinson's Disease Rating Scale, max. score of 199 points indicates the worst outcome
Change in disease severity measured by Hoehn & Yahr | Change from Baseline UPDRS at 12 months
  Hoehn & Yahr is a simple scale that describes disease severity on a scale of 0-5, with 5 indicating severe disability
Change in mobility, measured by Schwab- & England-Scale | Change from Baseline Schwab-&England-Scale at 12 months
  Schwab- & England-Scale assesses the capabilities of people with impaired mobility. The scale uses percentages with 100% indicating full independence.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Münster, Klinik für Neurologie, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Achtert K, Huchtemann T, Altendorf M, Kerkemeyer L, Haring M, Lummer C, Frenz L, Becking T, Friedmann J, Mildner P, Schwarze K, Steinhaus L, Amelung V, Warnecke T. Design and implementation of ParkinsonAKTIV: an interventional study to evaluate the effectiveness of a novel online platform to guide quickcard-based treatment decisions. Neurol Res Pract. 2023 Jun 1;5(1):23. doi: 10.1186/s42466-023-00249-5. PMID 37259124